CLINICAL TRIAL: NCT01198613
Title: A Double-blind, Randomised, Placebo-controlled Study to Evaluate Two Doses of ToleroMune Ragweed in Ragweed Allergic Subjects Following Challenge With Ragweed Allergen in an Environmental Exposure Chamber
Brief Title: ToleroMune Ragweed Exposure Chamber Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Circassia Limited (Industry)
Collaborators: Adiga Life Sciences, Inc. (Industry); Cetero Research, San Antonio (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TR002
Record Dates: First submitted 2010-09-06; First posted 2010-09-10 (Estimated); Last update posted 2011-10-07 (Estimated); Status verified 2011-10

CONDITIONS: Ragweed Allergy
Keywords: Ragweed allergy; Rhinoconjunctivitis; Exposure chamber; Immunotherapy; ToleroMune Ragweed

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Placebo (Placebo Comparator)
  Interventions: Biological: Placebo
- ToleroMune Ragweed Regimen 1 (Experimental)
  Interventions: Biological: ToleroMune Ragweed
- ToleroMune Ragweed Regimen 2 (Experimental)
  Interventions: Biological: ToleroMune Ragweed
- ToleroMune Ragweed Regimen 3 (Experimental)
  Interventions: Biological: ToleroMune Ragweed
- ToleroMune Ragweed Regimen 4 (Experimental)
  Interventions: Biological: ToleroMune Ragweed

INTERVENTIONS:
Biological: ToleroMune Ragweed — Intradermal injection 1 x8 administrations 2 weeks apart
  Arms: ToleroMune Ragweed Regimen 1; ToleroMune Ragweed Regimen 2; ToleroMune Ragweed Regimen 3; ToleroMune Ragweed Regimen 4
Biological: Placebo — Intradermal injection, 1x8 administrations 2 weeks apart
  Arms: Placebo

SUMMARY:
It is believe that ragweed is the primary cause of autumn allergies and 87% of patients with ragweed allergy suffer rhinoconjunctivitis. ToleroMune Ragweed is a novel, synthetic, allergen-derived peptide desensitising vaccine, currently being developed for the treatment of ragweed allergy.

This study will look at the efficacy, safety and tolerability of two doses of ToleroMune Ragweed in ragweed allergic subjects following challenge with ragweed in an EEC.

DETAILED DESCRIPTION:
This study is designed as a randomised, double-blind, placebo-controlled, parallel group study to evaluate the safety and tolerability of ToleroMune Ragweed in ragweed allergic subjects with allergic rhinoconjunctivitis,subjects may also have controlled asthma. The efficacy of ToleroMune Ragweed will be explored in subjects using an(Environmental Exposure Chamber)EEC.

The study will consist of 3 study periods. In Period 1, Screening will be performed up to a maximum of 12 weeks before randomisation and may consist of one or two visits to the clinic, at the Investigator's discretion. Baseline Challenge will consist of 4 visits to the EEC at least 3 days before randomisation.

In Period 2, subjects in each cohort complying with the inclusion/exclusion criteria will be randomised to one of five groups and will receive treatment every 2 weeks (±2 days) for 14 weeks.

In Period 3, Post Treatment Challenge will consist of 4 visits to the EEC 18-22 weeks after the first administration in the treatment period and assessments will be performed identical to those at the baseline challenge. Follow-up will be conducted 3-10 days after PTC.

ELIGIBILITY:
Inclusion criteria

* Male or female, aged 18-65 years.
* Minimum 2-year documented history of rhinoconjunctivitis on exposure to ragweed. [Subjects may also have controlled asthma
* Positive skin prick test to ragweed allergen.
* Minimum qualifying rhinoconjunctivitis symptom scores

Exclusion criteria

* History of asthma.
* A history of anaphylaxis to ragweed allergen.
* Subjects with an FEV1 <70% of predicted.
* Subjects who cannot tolerate baseline challenge in the EEC.
* Subjects for whom administration of epinephrine is contra-indicated (e.g. subjects with acute or chronic symptomatic coronary heart disease or severe hypertension).
* A history of severe drug allergy, severe angioedema or anaphylactic reaction to food.
* A history of any significant disease or disorder (e.g. cardiovascular, pulmonary, gastrointestinal, liver, renal, neurological, musculoskeletal, endocrine, metabolic, neoplastic/malignant, psychiatric, major physical impairment).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 275 (Estimated)
Dates: Start 2010-09; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Total Rhinoconjunctivitis Symptom Score | Upto 22 weeks

SECONDARY OUTCOMES:
Symptom scores for ocular and nasal symptoms | Upto 22 weeks
Acoustic Rhinometry | Upto 22 weeks
Skin prick testing | Baseline and final follow up
Ragweed specific IgE | At baseline and at follow up
Ragweed specific IgA | At baseline and follow up
Ragweed specific IgG4 | At baseline and at follow up
Adverse Events | Upto 23 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Deepen Patel, MD, CCFP, Principal Investigator — Cetero Research, San Antonio
Locations (2):
- Canada (2):
  - KGK Synergize Inc., London, Ontario
  - Cetero Research, Mississauga, Ontario